CLINICAL TRIAL: NCT05183698
Title: Spectroscopic Assessment of Autofluorescent Signatures of Tissue in and Around Wounds Identified by MolecuLight i:X Imaging Device
Brief Title: Point-spectroscopy Trial
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-002
Record Dates: First submitted 2021-12-07; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Wound; Wound of Skin
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Evaluation and characterization of autofluorescence signals of tissue in and around wounds as identified by MolecuLight fluorescence image.

DETAILED DESCRIPTION:
Evaluate and characterize autofluorescence signals of tissue components in and around wounds identified by MolecuLight FL images using a point spectrometer. The fluorescence spectroscopy data will yield quantitative spectral information, including the relative intensity and emission peak of the biological autofluorescence signatures.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute or chronic wounds
* 18 years or older
* Willing to consent

Exclusion Criteria:

* Treatment with an investigational drug within 1 month of enrolment
* Any contra-indication to regular wound care
* Inability or unwillingness to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic and/or acute wound
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2022-05-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Spectra of autofluorescent signatures of tissue in and around the wounds | 2 months
  Spectral characterization (i.e. emission curve including intensity) of the autofluorescence signal from wound tissue and surrounding tissue will be catalogued from all 50 study participants.